CLINICAL TRIAL: NCT06261723
Title: Effect of Non-chirurgical Periodontal Treatment on the Innate and Adaptive Immunity From a Gender Perspective: Potential Therapeutic Implications of microRNAs
Brief Title: Effect of Non-chirurgical Periodontal Treatment on the Immune System From a Gender Perspective
Status: Completed | Type: Observational
Sponsor: Milagros Rocha Barajas (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor-Investigator, Milagros Rocha Barajas, Senior Postdoctoral Researcher, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Organization: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Other Study IDs: PI22/1009
Record Dates: First submitted 2024-01-30; First posted 2024-02-15 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Periodontal Diseases
Keywords: inflammation; atherosclerosis; gingivitis; oxidative stress; Obesity
MeSH Terms: conditions — Periodontal Diseases; Inflammation; Atherosclerosis; Gingivitis; Obesity | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group without obesity: Control Group with periodontitis and without obesity
  Interventions: Procedure: non-chirurgical periodontal treatment
- Obesity Group: Obesity Group with periodontitis
  Interventions: Procedure: non-chirurgical periodontal treatment

INTERVENTIONS:
Procedure: non-chirurgical periodontal treatment — The non-chirurgical periodontal treatment (scaling and root planing) is the gold standard procedure in therapy for periodontitis. It involves the mechanical removal of plaque and bacterial deposits, creating a local microbial environment in harmony with periodontal health and promoting the replacement of damaged periodontal tissues with collagen-rich connective tissues. This favors a shift in the composition of the oral microbiota from a community dominated by Gram-negatives to one dominated by Gram-positives.
  Other Names: scaling and root planing

SUMMARY:
The goal of this observational study is to evaluate non-surgical periodontal treatment in women and men with periodontitis with and without obesity. The main questions it aims to answer are:

* If non-surgical periodontal treatment of patients with chronic periodontitis can modulate the innate and adaptive immune response taking into account patient gender and the coexistence of obesity
* If there are specific miRNAs that can regulate this immune response and can be considered as suitable biomarkers and therapeutic targets.

Obese or non-obese participants with periodontitis will receive non-surgical periodontal treatment, consisting of oral health guidance and mechanical periodontal debridement throughout the mouth using an ultrasonic device and manual curettes. Researchers will compare four groups: obese women, non-obese women, obese men, and non-obese men, to clarify the involment of immune response after treatment, considering the coexistence of obesity and potential gender differences.

DETAILED DESCRIPTION:
Blood, gingival crevicular fluid (GCF), and saliva samples will be collected from patients at baseline and 12 weeks after non-surgical periodontal treatment. From fasting blood samples (12h), peripheral blood mononuclear cells (PBMCs) and neutrophil fractions will be isolated using an immunomagnetic method, following the manufacturer's protocol, and plasma and serum will be stored at -80°C until analysis. LUNA-FL will be used to determine cell count and viability (acridine orange and propidium iodide double stain) in cell samples. GCF samples will be collected in duplicate by carefully inserting sterile paper points into the periodontal pocket 1 mm for 30 s. The volume will be determined using the Periotron 8000 and stored at -80°C for future determinations. Unstimulated saliva will be collected in RNase-free tubes by expectoration, and after centrifugation, the supernatant will be stored at -80°C for microRNA (miRNA) analysis.

Clinical periodontal parameters of probing pockets depth (PD), millimetres of clinical attachment level (CAL), bleeding on probing (BOP), simplified plaque index of Silness and Löe, and simplified calculus index of Greene and Vermillion will be determined using a conventional manual periodontal probe (UNC-15 PCP). A periodontal examination will be performed to measure PD, CAL, and BOP at six sites per tooth for all teeth, excluding third molars, as previously described. Patients will be interviewed about their medical history, lifestyle habits (smoking, frequency of tooth brushing, physical activity), and sociodemographic characteristics. Weight, height, and blood pressure will be measured using standardized methods. Biochemical parameters of carbohydrate metabolism - glucose, insulin, glycated hemoglobin (A1c) -, lipid profile - total cholesterol, LDL, HDL, triglycerides (TG), apolipoproteins AI and B -, emerging inflammatory and cardiovascular risk markers - C-Reactive Protein (CRP), C3c, and retinol-binding protein 4 (RBP4) -, and complete blood count will be determined at the hospital's Clinical Analysis Service.

For detection of differences in protein expression, cells will be incubated in lysis buffer with protease and phosphatase inhibitors (RIPA Buffer) for 15 minutes at 4 degrees celsius (°C). The supernatant will be collected after centrifugation for 15 minutes at 16,000g. The total protein concentration will be quantified using a bicinchoninic acid (BCA) protein assay. Aliquots of 25 µg of protein will be resolved on 8-16% gradient SDS-polyacrylamide gels and transferred to nitrocellulose membranes. Target proteins will be detected by incubating the membranes with anti-actin, JNK, NFkB, MCP1, GPX-1, NLRP3, ASC, procaspase 1, caspase 1, NADPH oxidase, catalase, GPX1, SOD1, Beclin, ATG5-ATG12, p62, LC3 I, LC3 II, Pink1, GRP78, eIF2alpha, IRE1 alpha, ATF6, CHOP, PGC1 alpha, mTFA, VDAC, Complex I, II, III, IV and V. The protein signal will be detected by chemiluminescence and analyzed by densitometry.

Inflammasome complex assembly (first stage of activation) through co-localization studies of NLRP3-ASC in PBMCs will be conducted using the confocal and/or fluorescence microscopy. Briefly, PBMCs will be seeded on coverslips coated with Poly-D-Lysine, fixed with paraformaldehyde (PFA) 4% for 20 minutes, permeabilized with Triton X-100 for 20 minutes and blocking with Phosphate-buffered saline buffer-Bovine serum albumn (PBS-BSA) 3% for 1 hour at room temperature. Hybridization with specific primary antibodies (diluted in PBS-BSA 1%) will be carry out overnight at 4 ºC and then, secondary antibodies conjugated with AlexaFluor fluorophores will be incubated for 1 hour in the dark at room temperature. Stained samples will be transferred the coverslip onto microscope slide and conserved in anti-fade fluorescence mounting medium.

Circulating levels of cytokines, adhesion molecules and serum oxidative stress markers will be measured in serum samples, but for secretome studies 1x10^6 PBMCs will be previously incubated in 1 mL RPMI with 10% fetal bovine serum (FBS) for 4 hours (37°C, 5% CO2) to obtain the supernatant. Both serums and supernatants will be analyzed with a Luminex® 200 analyzer system following the Milliplex® MAP Kit manufacturer's procedure. These same determinations will be carried out on GCF and serum/plasma samples from patients.

The quantification of functional autophagosomes in PBMCs will be performed using flow cytometry on our BD Accuri equipment with the CYTO-ID® Autophagy detection kit following manufacturer's procedure. In parallel, leucocyte from whole blood samples will be incubated with redox status detecting fluorescent probes for 15 minutes and then, they will be analysed using flow cytometry. Additionally, a multicolor panels for flow cytometry based on cluster of differentiation (CD) antigens detection, CD3/CD4/CD8/CD45RA/CCR7/CD38 and CD14/CD16, will be designed to analyze the percentage of lymphocyte T subpopulations (naive T cells (TN), central memory (TCM), effector memory (TEM) and terminally differentiated (TEMRA) cells) and, monocytes subpopulations (classical, non-classical, and intermediate), respectively in blood samples. In both procedures 10000 events will be acquired and single staining and FMO controls for all fluorochrome-conjugated antibodies in the panels will be performed to establish adequate compensation and define positive signals.

A parallel plate flow chamber, connected to an inverted microscope, will enable the researchers to measure neutrophil-endothelial cell interactions in vitro. Through this system, the leukocyte suspension obtained from patients will be perfused over a monolayer of immortalized endothelial cells (HUVEC/TERT 2) under conditions simulating blood flow. Videos will be analyzed afterward to determine flow, rolling velocity, and firm adhesion of leukocytes to endothelial cells, as previously described (Antioxidants. 2020 Aug 11;9(8):734).

Changes in gene expression levels will be evaluated using Nanostring® technology for nCounter®. To sum up, total RNA will be extracted from PBMCs using the GeneAllR RibospinTM total kit, and starting from 100-200 ng of total RNA, Diagnostica Longwood, S.L. will analyze the differential gene expression response, thus obtaining the multiplex metabolism panel.

For differential gene expression analysis of miRNAs (DEGs), RNA will be extracted using the miRNeasy Serum/Plasma kit (Qiagen). After short-chain RNA extraction, libraries will be prepared for sequencing using the TruSeq Small RNA library preparation kit (Illumina, Inc). Libraries will be pooled equimolarly and quantified using the KAPA SYBR FAST Universal qPCR kit with Illumina Primer Premix, and group size will be measured using a Bioanalyzer (Agilent). Finally, 2 nanomoles of the group will be sequenced on the Illumina NovaSeq6000 platform with a 1% PhiX control in the FISABIO facilities. Libraries will be sequenced using 2x100 bp chemistry in an SP flow cell (Illumina, Inc). After multiplexing, raw data will be processed using the "COMPSRA: a COMprehensive Platform for Small RNA-Seq data Analysis" pipeline.

DNA will also be extracted from plasma according to the "blood and body fluid protocol" of the QIAamp blood reagent set (QIAgen, Hilden, Germany); 400 μL of plasma will be applied to each column, DNA will be eluted in 200 μL of supplied buffer and will be stored at -20°C until use. mtDNA will be quantified with reverse transcription-quantitative polymerase chain reaction (RT-qPCR) using specific primers for obtaining circulating mtDNA levels.

Data analysis will be performed with SPSS 17.0. Groups will be compared using unpaired Student's t-tests or Mann-Whitney U tests for parametric and non-parametric data, respectively. Changes after intervention will be evaluated using paired Student's t-tests or Wilcoxon tests, depending on the variable distribution. Pearson or Spearman correlation coefficients will be used to measure the strength of association between variables. In multivariable regression models, the relationship between two or more explanatory variables (independent variables) and a response variable (dependent variable) will be evaluated by fitting a linear equation to the obtained data. Qualitative data will be expressed in percentages, and proportions will be compared using a Chi-square test. All tests will use a 95% confidence interval, and differences will be considered statistically significant when p <0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Men/Women with periodontitis:

   * Periodontitis will be diagnosed according to the definition of the Centers for Disease Control and Prevention / American Academy of Periodontology (CDC/AAP).
2. Men/Women with obesity:

   * Body mass index (BMI) ≥30 kg/m2 (WHO 2000)

Exclusion Criteria:

* Having fewer than fourteen teeth,
* Having infectious diseases
* Having other oral inflammatory diseases,
* Having received periodontal treatment in the past six months or antibiotics in the previous three months, undergoing systemic anti-inflammatory treatment,
* Pregnancy or lactation
* Serious illnesses, congenital adrenal hyperplasia, virilizing tumors, hypothyroidism, Cushing's syndrome, prolactinomas, cardiovascular diseases, or diabetes mellitus.
* Alcohol or drug abuse
* Psychiatric disorders.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — According to presence of periodontitis and obesity.
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Changes in inflammasome complex activation grade in patients with chronic periodontitis with and without obesity, before and after non-surgical periodontal treatment. | At recruitment
  Relative protein expression of NLRP3, ASC, Caspase-1, AIM2, IL-1β, IL-18 and inflammatory mediators NFκB, JNK, IL6, and TNFα by Western Blot and normalized to the loading control protein, and inflammasome assembly by confocal microscopy in PBMC.
Changes in endothelial function in the study population. | At recruitment
  Evaluation of leucocytes adhesion to the endothelial cell in vitro by means of a parallel flow chamber system coupled to an inverted phase-contrast microscope.
Changes in endothelial function at molecular level in the study population. | At recruitment
  Evaluation of circulating levels of adhesion molecules - P-selectin, ICAM-1, and VCAM-1, and circulating cytokines (L1β, IL18, IL6 and TNFα) in serum using Luminex technique.
Changes in the systemic inflammation status in the study population. | At recruitment
  Evaluation of circulating levels of mtDNA in plasma samples using RT-PCR.
Changes in the expression of genes related to inflammatory pathways in PBMC in the study population. | At recruitment
  Relative expression of genes related to inflammatory pathways (TLR and NFkB) by means of nanostring technology.
Changes in the expression of genes related to oxidative stress levels in PBMC in the study population. | At recruitment
  Relative expression of genes related to oxidative stress (GSR, GPX1, GPX2, SOD, CAT, TXNRD1, AKR1B10, SLC7A11, GCLC, GCLM) by means of nanostring technology.
Changes in the expression of genes related to cellular respiration in PBMC in the study population. | At recruitment
  Relative expression of genes related to mitochondrial respiration (I, II, III, IV and V complexes) in PBMC by means of nanostring technology
Sequence miRNAs in biological fluids in patients with chronic periodontitis with and without obesity, before and after non-surgical periodontal treatment. | At recruitment
  Analysis of differential gen expression (DEGs) of miRNAs
Evaluate the distribution and phenotype of different T lymphocyte and monocyte subpopulations in the study population. | At recruitment
  Detection of T lymphocyte subpopulations with CD3/CD4/CD8/CD45RA/CCR7/CD38 multicolor panel and monocyte subpopulations with CD14/CD16 multicolor panel by flux cytometry.

SECONDARY OUTCOMES:
Changes in the protein expression of autophagy markers in PBMC in the study population. | At recruitment
  Relative expression of intracellular proteins related to autophagy/mitophagy mechanisms (Beclin 1, ATG5, LC3II/I, p62, NRB1, PINK1, MIEAP) assessed by western blot and normalized to the loading control protein.
Evaluate autophagy flux in the study population. | At recruitment
  Quantification of cationic amphiphilic tracer (CAT) probe which label vacuoles associated with the autophagy pathway by flux cytometry in PBMC.
Evaluate autophagosome formation in the study population. | At recruitment
  Detection of LC3 puntae by confocal/fluorescence microscope in PBMCs.

CONTACTS AND LOCATIONS:
Overall Officials: Milagros Rocha, PhD, Principal Investigator — FISABIO-HOSPITAL DR PESET
Locations (2):
- Spain (2):
  - University Hospital Dr Peset, Valencia, Valencia
  - University Hospital Dr. Peset, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fruhbeck G. Obesity: Screening for the evident in obesity. Nat Rev Endocrinol. 2012 Oct;8(10):570-2. doi: 10.1038/nrendo.2012.165. Epub 2012 Sep 4. No abstract available. PMID 22945363
- [Background] Rocha VZ, Libby P. Obesity, inflammation, and atherosclerosis. Nat Rev Cardiol. 2009 Jun;6(6):399-409. doi: 10.1038/nrcardio.2009.55. Epub 2009 Apr 28. PMID 19399028
- [Background] Tonetti MS. Periodontitis and risk for atherosclerosis: an update on intervention trials. J Clin Periodontol. 2009 Jul;36 Suppl 10:15-9. doi: 10.1111/j.1600-051X.2009.01417.x. PMID 19432627
- [Background] Virto L, Cano P, Jimenez-Ortega V, Fernandez-Mateos P, Gonzalez J, Esquifino AI, Sanz M. Obesity and periodontitis: An experimental study to evaluate periodontal and systemic effects of comorbidity. J Periodontol. 2018 Feb;89(2):176-185. doi: 10.1902/jop.2017.170355. Epub 2018 Feb 16. PMID 28914596
- [Background] Isaza-Guzman DM, Medina-Piedrahita VM, Gutierrez-Henao C, Tobon-Arroyave SI. Salivary Levels of NLRP3 Inflammasome-Related Proteins as Potential Biomarkers of Periodontal Clinical Status. J Periodontol. 2017 Dec;88(12):1329-1338. doi: 10.1902/jop.2017.170244. Epub 2017 Jul 10. PMID 28691886
- [Background] Trexler M, Patthy L. Residues Cys-1 and Cys-79 are not essential for refolding of reduced-denatured kringle 4 fragment of human plasminogen. Biochim Biophys Acta. 1984 Jun 28;787(3):275-80. doi: 10.1016/0167-4838(84)90320-0. PMID 6329306
- [Background] Moura MF, Navarro TP, Silva TA, Cota LOM, Soares Dutra Oliveira AM, Costa FO. Periodontitis and Endothelial Dysfunction: Periodontal Clinical Parameters and Levels of Salivary Markers Interleukin-1beta, Tumor Necrosis Factor-alpha, Matrix Metalloproteinase-2, Tissue Inhibitor of Metalloproteinases-2 Complex, and Nitric Oxide. J Periodontol. 2017 Aug;88(8):778-787. doi: 10.1902/jop.2017.170023. Epub 2017 May 11. PMID 28492359
- [Background] Martinez-Herrera M, Lopez-Domenech S, Silvestre FJ, Silvestre-Rangil J, Banuls C, Victor VM, Rocha M. Chronic periodontitis impairs polymorphonuclear leucocyte-endothelium cell interactions and oxidative stress in humans. J Clin Periodontol. 2018 Dec;45(12):1429-1439. doi: 10.1111/jcpe.13027. Epub 2018 Nov 20. PMID 30362144
- [Background] Chapple IL, Matthews JB. The role of reactive oxygen and antioxidant species in periodontal tissue destruction. Periodontol 2000. 2007;43:160-232. doi: 10.1111/j.1600-0757.2006.00178.x. No abstract available. PMID 17214840
- [Background] Kanzaki H, Wada S, Narimiya T, Yamaguchi Y, Katsumata Y, Itohiya K, Fukaya S, Miyamoto Y, Nakamura Y. Pathways that Regulate ROS Scavenging Enzymes, and Their Role in Defense Against Tissue Destruction in Periodontitis. Front Physiol. 2017 May 30;8:351. doi: 10.3389/fphys.2017.00351. eCollection 2017. PMID 28611683
- [Background] Park MH, Jeong SY, Na HS, Chung J. Porphyromonas gingivalis induces autophagy in THP-1-derived macrophages. Mol Oral Microbiol. 2017 Feb;32(1):48-59. doi: 10.1111/omi.12153. Epub 2016 Feb 24. PMID 26792079
- [Background] Tonetti MS, D'Aiuto F, Nibali L, Donald A, Storry C, Parkar M, Suvan J, Hingorani AD, Vallance P, Deanfield J. Treatment of periodontitis and endothelial function. N Engl J Med. 2007 Mar 1;356(9):911-20. doi: 10.1056/NEJMoa063186. PMID 17329698
- [Background] Luan X, Zhou X, Naqvi A, Francis M, Foyle D, Nares S, Diekwisch TGH. MicroRNAs and immunity in periodontal health and disease. Int J Oral Sci. 2018 Aug 6;10(3):24. doi: 10.1038/s41368-018-0025-y. PMID 30078842
- [Background] Yoneda T, Tomofuji T, Ekuni D, Azuma T, Maruyama T, Fujimori K, Sugiura Y, Morita M. Serum microRNAs and chronic periodontitis: A case-control study. Arch Oral Biol. 2019 May;101:57-63. doi: 10.1016/j.archoralbio.2019.03.009. Epub 2019 Mar 13. PMID 30889506